CLINICAL TRIAL: NCT00085787
Title: A Study of ARRY-142886 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRY-0401
Record Dates: First submitted 2004-06-14; First posted 2004-06-17 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — AZD 6244

ARMS (1):
- ARRY-142886 (Experimental)
  Interventions: Drug: ARRY-142886, MEK inhibitor; oral

INTERVENTIONS:
Drug: ARRY-142886, MEK inhibitor; oral — Part 1: single dose and multiple dose, escalating; Part 2: multiple dose, single schedule

SUMMARY:
This is a Phase 1 study during which patients with advanced solid tumors will receive investigational study drug ARRY-142886.

This study has 2 parts. In the first part, patients will receive increasing doses of study drug in order to achieve the highest dose of study drug possible that will not cause unacceptable side effects. Approximately 25 patients from the US will be enrolled in Part 1 (Completed).

In the second part of the study, patients will receive the best dose of study drug, determined from the first part of the study, and will be followed to see what side effects the study drug causes and what effectiveness the study drug has, if any, in treating the cancer. Approximately 35 patients from the US will be enrolled in Part 2 (Completed).

ELIGIBILITY:
Key Inclusion Criteria (Part 2):

* Histopathologically or cytologically confirmed solid tumor that is refractory to standard therapies, or for which no standard therapies exist, or for which the Investigator feels no other active therapy is required for the duration of the study.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Estimated life expectancy of greater than or equal to 3 months.
* Patient must have a tumor that is accessible for biopsy and must consent to paired tumor biopsies and normal skin biopsies being taken pre- and post-dose of study drug.
* Additional criteria exist.

Key Exclusion Criteria (Part 2):

* Uncontrolled or symptomatic brain metastases.
* Use of investigational drug or device within 30 days prior to first dose of study drug.
* Major surgery within 30 days prior to study start.
* Radiotherapy or chemotherapy within 21 days prior to study start (not including palliative radiotherapy at focal sites).
* Pregnancy or lactation.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-06; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | Part 1
Establish the maximum tolerated dose (MTD) of study drug. | Part 1
Assess the biological activity of the study drug in tumors in terms of inhibition of extracellular signal-regulated kinase (ERK) phosphorylation. | Part 2

SECONDARY OUTCOMES:
Characterize the pharmacokinetics (PK) of the study drug in terms of plasma concentrations. | Part 1 and Part 2
Characterize the pharmacodynamic (PD) activity of the study drug on biomarkers. | Part 1 and Part 2
Assess the efficacy of the study drug in terms of tumor dimension assessment. | Part 1 and Part 2
Confirm the safety of the study drug at the MTD as determined by adverse events, clinical laboratory tests, vital signs and electrocardiograms. | Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Anschutz Cancer Center, Aurora, Colorado
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania